CLINICAL TRIAL: NCT06284759
Title: The Effect of Tele-Nursing Application Based on Orem's Self-Care Theory on Self-Care Ability and Daily Living Activities in Trauma-Related Lower Extremity Fracture Surgery Patients
Brief Title: The Effect of Tele-Nursing Application on Self-Care Ability and Daily Living Activities in Fracture Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Lokman Hekim University (Other Government); Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Sevil Güler, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-77082166-302.08.01-380534
Record Dates: First submitted 2024-02-09; First posted 2024-02-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Lower Extremity Fracture
Keywords: Activities of Daily Living; Orem's Self Care Theory; Trauma Nursing; Tele-nursing; Lower extremity fracture surgery; Self care agency; Orthopaedic and trauma nursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In the study, the statistician was blinded using the blind technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention group were monitored with a tele-nursing application based on Orem's Self-Care Theory, and training and counseling were provided for 6 weeks after discharge. Post-discharge interviews were conducted by resercher via phone call and video conference (zoom, WhatsApp, etc.). The video conference method was presented to the patient's preference and the decision was made together. The interview with each patient lasted an average of 30 minutes. Patients in the intervention group were sent infographics prepared in line with the theory, including the interview content and suggestions after each interview. The study focuses on post-discharge tele-nursing practice follow-up outcomes. Baseline data were collected at the hospital on the 2nd and 3rd postoperative day. Post-discharge data were collected on the 7th-10th day, 18th-21st day and 40th-45th day.
  Interventions: Other: post-discharge telenursing intervention
- Control (No Intervention): Patients in the control group were discharged in accordance with the current hospital procedure. No intervention was made. The study focuses on post-discharge tele-nursing practice follow-up outcomes. Baseline data were collected at the hospital on the 2nd and 3rd postoperative day. Post-discharge data were collected on the 7th-10th day, 18th-21st day and 40th-45th day. It was collected by phone call or video conference (zoom, WhatsApp, etc.).

INTERVENTIONS:
Other: post-discharge telenursing intervention — Tele-nursing based on Orem's Self-Care Theory was applied to patients with lower extremity fracture surgery. Phone/video calls 24-48 after discharge. hours, 7-10. day,18-21. day, 28-30th day and 40-45th day. day was made. Telephone or video conference interviews were held on the day and time convenient for the patient. After each meeting, the date and time of the next meeting was planned. The video conferencing method (zoom, skype, whatsapp, etc.) was presented to the patient's preference and the decision was made together. In phone/video conference calls, patients were informed about their current problems. Additionally, patients' questions were answered. Prior to tele-nursing monitoring, the researchers identified emergent or urgent situations; Patients were informed that they should consult their doctor if this occurs. The interview with each patient lasted an average of 30 minutes.
  Arms: Intervention

SUMMARY:
This study aims to determine the effect of tele-nursing application based on Orem's Self-care Theory on self-care agency and daily living activities in trauma-related lower extremity fracture surgery patients.

DETAILED DESCRIPTION:
The research was conducted to determine the effect of tele-nursing application based on Orem's Self-care Theory on self-care agency and daily living activities in trauma-related lower extremity fracture surgery patients. The research was planned as a randomized controlled experimental type study. 52 patients (intervention 26, control 26) were included in the study sample using the "simple randomization method". In order to collect the data, Introductory Information Form, Self-Care Agency Scale, KATZ Activities of Daily Living Scale and Lawton Brody Activities of Daily Living Scale were used. Current hospital procedures were applied to patients in the control group without any intervention. Patients in the intervention group were monitored with a tele-nursing application based on Orem's Self-Care Theory, and training and counseling were provided for 6 weeks after discharge. Data; It was collected face to face once before discharge in both groups, and three times by video conference method: 7-10 days, 18-21 days and 40-45 days after discharge. Tele-Nursing Application Monitoring Form and reminder infographics, prepared based on Orem's Self-Care Theory, were used in the follow-up process of patients who had trauma-related lower extremity fracture surgery. Chi square, independent samples t test, analysis of variance in repeated measurements and Pearson correlation analysis were used to analyze the data. While there was no statistical difference between the groups in the first measurements, in the 2nd, 3rd and 4th measurements, the intervention group's self-care agency, KATZ activities of daily living and Lawton Brody instrumental activities of daily living scale scores were found to be statistically significantly higher than the control group (p<0, 05). In this study, it was concluded that tele-nursing application based on Orem Self-Care Theory has a positive effect on self-care agency and daily life activities.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* Agreeing to participate in the study voluntarily,
* Able to understand and speak Turkish,
* At least primary school graduate,
* Those who have undergone lower extremity fracture surgery,

Exclusion Criteria:

* Over 65 years of age,
* Having an uncontrollable medical problem,
* Having a hip fracture or fragility fracture due to a fall,
* Having an external fixator,
* Amputation develops,
* People whose speech, hearing and visual disabilities prevent them from participating in telenursing monitoring will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Self Care, Assessed using the Self-Care Agency scale. | Baseline data were collected at the hospital on the 2nd and 3rd postoperative day. Post-discharge data were collected on the 7th-10th day, 18th-21st day and 40th-45th day.
  The scale is a 5-point Likert-type and each statement is scored from 0 to 4. Among the response options, 0 points are given to the answer "It doesn't describe me at all", 1 point is given to the others, respectively, "It doesn't describe me much", 2 points are given to "I have no idea", 3 points are given to the answer "It describes me a little" and 4 points are given to the answer "It describes me a lot". In the Turkish-translated scale, 8 items (items 3, 6, 9, 13, 19, 22, 26 and 31) are evaluated as negative and the scoring is reversed. The maximum score is 140. A high score from the scale indicates the high level of self-care or self-care ability and strength of the individual.
Activities of daily living, Assessed using the Katz index of independence in activities of daily living (ADL) scale. | Baseline data were collected at the hospital on the 2nd and 3rd postoperative day. Post-discharge data were collected on the 7th-10th day, 18th-21st day and 40th-45th day.
  The scale measures the degree of addiction in self-care activities, which consists of six headings: bathing, dressing, toilet needs, mobility, excretion and nutrition. The total score from the scale varies between 0-6. A low score indicates a high level of addiction. According to the results of the Katz Activities of Daily Living Scale, 0-2 points are classified as dependent, 3-4 points are classified as semi-dependent, and 5-6 points are classified as independent.
Instrumental activities of daily living, Assessed using the The Lawton instrumental activities of daily living scale. | Baseline data were collected at the hospital on the 2nd and 3rd postoperative day. Post-discharge data were collected on the 7th-10th day, 18th-21st day and 40th-45th day.
  The scale consists of a total of 8 items and a single sub-dimension, including the ability to use the phone, shopping, meal preparation, house cleaning, laundry, travel, responsibility for taking medications, and financial affairs. The total score from the scale varies between 0-8. A low score indicates a high level of addiction.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No